CLINICAL TRIAL: NCT02028325
Title: Yellow 560 Microscope for Intraoperative Visualization of Fluorescein Stained Intracranial Lesions
Acronym: Fluorescein
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment. No new subjects had been enrolled for nearly a year.
Sponsor: Indiana University (Other)
Collaborators: Sentara Norfolk General Hospital (Other)
Responsible Party: Principal Investigator, Aaron Cohen-Gadol, Neurosurgeon, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCBS-0003
Record Dates: First submitted 2013-12-18; First posted 2014-01-07 (Estimated); Results first posted 2016-09-29 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-10

CONDITIONS: Adult Intracranial Neoplasm; Vascular: Intracranial
MeSH Terms: conditions — Brain Neoplasms | interventions — Fluorescein; Fluoresceins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluorescein Sodium (Experimental): All patients enrolled in the study will prepare for surgery as per standard neurosurgical indications, procedures and institution protocols. At the time of the anesthesia induction, with the patient under general anesthesia, Fluorescein Sodium 10% (100mg/1mL) at a dose of 3-20 mg/kg will be administered intravenously (the optimal dosage will be determined within the study as the most minimal dose for adequate visualization will be used). For vascular lesions, fluorescein sodium 10% (100mg/1mL) will be injected and used to assess its application after the conventional methods have confirmed the exclusion of the aneurysm. No patient's care will be affected by the results of the Fluorescein angiography.
  Interventions: Drug: Fluorescein Sodium

INTERVENTIONS:
Drug: Fluorescein Sodium — All patients enrolled in the study will prepare for surgery as per standard neurosurgical indications, procedures and institution protocols. At the time of the anesthesia induction, with the patient under general anesthesia, Fluorescein Sodium 10% (100mg/1mL) at a dose of 3-20 mg/kg will be administered intravenously (the optimal dosage will be determined within the study as the most minimal dose for adequate visualization will be used). For vascular lesions, fluorescein sodium 10% (100mg/1mL) will be injected and used to assess its application after the conventional methods have confirmed the exclusion of the aneurysm. No patient's care will be affected by the results of the Fluorescein angiography.
  Other Names: AK-Fluor

SUMMARY:
The purpose of this study is to evaluate the effectiveness of using Fluorescein Sodium and the Yellow 560 microscope to aid in treatment of intracranial tumors and vascular lesions.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of using Fluorescein Sodium and the Yellow 560 microscope to aid in treatment of intracranial tumors and vascular lesions. The objectives of this study aim to investigate the use of Fluorescein in assisting with evaluating complete tumor removal and thorough treatment of intracranial vascular lesions as well as tumor biopsy procedures. The hypothesis is that Fluorescein Sodium will help surgeons better identify residual tumor and vascular lesions and its use will allow surgeons to obtain better surgical results and prognostic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Diagnosed by preoperative imaging modalities to have a brain tumor or vascular lesions (aneurysm, arteriovenous malformation or arteriovenous fistula) requiring surgical intervention.
* The patient is determined by a board certified Neurosurgeon (above mentioned neurosurgeons) to benefit from the application of Fluorescein Sodium intraoperatively
* Patient or legally authorized representative provides written informed consent to enroll in this study.

Exclusion Criteria:

* Known allergic reaction to Fluorescein Sodium.
* Children.
* Prisoners.
* Students.
* Infection of the central nervous system or other sites.
* Hemodynamic instability or significant impairments in circulation.
* Concomitant treatment with other investigational drugs.
* Any uncontrolled condition unrelated to the neurosurgical disease.
* History of psychiatric, additive, or any other disorder that compromises the ability to provide informed consent or comply with study protocols.
* Participation on other clinical trials during the last thirty days.
* Pregnant patients.
* Patients unable to discontinue medications that affect Fluorescein metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron A Cohen, MD, MSc, Principal Investigator — IU Health Methodist Hospital
Locations (2):
- United States (2):
  - Aaron Cohen-Gadol, MD, Indianapolis, Indiana
  - Sentara Norfolk General Hospital, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants failed screening
Period: Overall Study
Arm/Group | Fluorescein Sodium
Started | 136
Completed | 126
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Fluorescein Sodium
Number analyzed (Participants) | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 104
  >=65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 64

OUTCOME MEASURES:

1. Primary Outcome: Concordance Between Surgical Impression of Residual Lesion and Appearance on Post-operative Imaging
Description: We will perform fluorescein fluorescence/angiography at surgery and assess if fluorescence reveals any residual tumor or vascular lesion (aneurysm, arteriovenous malformation, or arteriovenous fistula) following surgical intervention. For subjects with brain tumors we will then perform a regular postoperative MRI and assess if there was any residual tumor and measure the accuracy of fluorescein fluorescence to assess the amount of the residual tumor seen on the postoperative MRI. Similarly, for the aneurysms or other vascular lesions, we will perform a regular postoperative angiogram and assess the accuracy of fluorescein angiography results in estimating the amount of residual lesion.
Time Frame: up to 1 week. For subjects where clinical post-operative MRI/angiography was not performed within 7 days, MRI/angiography completed within 3 months post-operatively was utilized for evaluation.
Measure: Number; unit: participants
Arm/Group | Fluorescein Sodium
Number analyzed (Participants) | 126
participants
  Concordance | 84
  Nonconcordance | 10
  Unable to reliably assess | 32

ADVERSE EVENTS:
Arm/Group | Fluorescein Sodium
Serious Adverse Events (participants affected / at risk) | 0/126
Other Adverse Events (participants affected / at risk) | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No